CLINICAL TRIAL: NCT07319923
Title: Establishment and Promotion of an AI-Based Early Warning System for Prostate and Bladder Cancer Screening in the Male Community Population of Beijing
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BJCP-AI-UroScreen-2025-001
Record Dates: First submitted 2025-12-20; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer; Community-based Screening
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Prostate cancer is one of the most common malignancies in the male genitourinary system, and it is also the cancer with the fastest-growing incidence and mortality rates among men in China. Although prostate cancer screening can significantly reduce mortality, China has not yet established a well-developed screening system, which is one of the reasons why its mortality rate remains notably higher than that of Western countries. The primary objective of this project is to establish an efficient screening-diagnosis-treatment pathway, beginning with screening in community hospitals, followed by definitive diagnosis in secondary hospitals, and finally treatment in tertiary hospitals. Additionally, the project aims to achieve multi-institutional and multi-terminal sharing of disease information as well as dynamic monitoring and follow-up. The feasibility and effectiveness of this model will be validated through statistical analysis of the data.

ELIGIBILITY:
Inclusion Criteria:

* Male community residents aged 50 years or older;

Life expectancy > 10 years and ECOG performance status of 0-2;

Permanent residents of Beijing who are willing to cooperate with researchers in the screening process, complete required tests and questionnaires, and participate in subsequent follow-up;

Support for the research project and provision of signed informed consent.

Exclusion Criteria:

* 1）Presence of any other malignant tumor or pre-existing prostate malignancy; 2）Presence of prostatitis or active infection in other parts of the urinary system; 3）Inability to cooperate with the study procedures or other factors deemed unsuitable for participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study targets male community residents aged 50 years or above who can actively cooperate with researchers in the screening process by completing relevant procedures such as urine and blood sample collection.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Serum PSA level | from 2025 to 2027

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Peking University First Hospital, Beijing, 100034, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes